CLINICAL TRIAL: NCT05095870
Title: Evaluation of the Peripheral Nerve Ultrasound as a Diagnostic Tool in CANVAS (Cerebellar Ataxia With Neuropathy and Vestibular Areflexia Syndrome) Neuronopathies
Brief Title: Evaluation of the Peripheral Nerve Ultrasound as a Diagnostic Tool in CANVAS Neuropathies
Acronym: CANVAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/II-02
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-05

CONDITIONS: Neuropathy; Cerebellar Ataxia; Neurodegenerative Diseases
MeSH Terms: conditions — Cerebellar Ataxia; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CANVAS Patients: Patient with a CANVAS diagnosis with genetic evidence (RFC1+)
  Interventions: Other: No intervention
- control group: Patient with axonal sensory-motor or pure sensitive neuropathy confirmed by electroneuromyography
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Pure observational study

SUMMARY:
Cerebellar ataxia with neuropathy and bilateral areflexia syndrome (CANVAS) is a late onset neurodegenerative disorder with a slowly progressive ataxia. It's genetic causative etiology with an autosomal recessive inheritance has a recent discovery.

It is clinically characterized by impaired visually enhanced vestibulo-ocular reflex, although patients commonly present with imbalance as a main concern, associated with sensory complaints. It has been demonstrated that sensory impairment in CANVAS patients is due to degeneration of dorsal root with abnormal sensory nerve conduction.

Previously defined diagnostic criteria included cerebellar atrophy on brain MRI, neuronopathy on electrophysiological studies and negative genetic testing for other inherited ataxia syndromes like Friedriech ataxia and spinal cerebellar ataxia (SCA).

Peripheral nerve ultrasound is a noninvasive technique, able to identify abnormal peripheral nerves with underlying injuries and specific sonographic characteristics. Pelosi et al established that patients with CANVAS have a smaller nerve cross sectional area (CSA) compared to healthy individuals and/ or axonal neuropathies.

The main objective of this study was to obtaine a detailed description of peripheral nerves in consecutive patients with CANVAS syndrome followed in theneurology department of the Universitary Hospital of Nimes (France), using conventional electrophysiology and peripheral nerve ultrasound.

ELIGIBILITY:
CANVAS Patients :

Inclusion Criteria:

* Patients followed at the University Hospital of Nîmes between 2018-2021
* Age > 18 years
* Diagnosis of CANVAS with genetic evidence (RFC1+)
* Diagnosis of neuronopathy

Exclusion Criteria:

* Age <18 years
* Chronic polyradiculoneuritis or other demyelinating neuropathy

Control group, inclusion criteria :

Patient with axonal sensory-motor or pure sensory neuropathy confirmed by electro neuromyography, and concordant with the clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with CANVAS syndrome followed in our neurology department, using conventional electrophysiology and peripheral nerve ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
median ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of median nerve ultrasound
ulnar nerve at wrist ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of ulnar nerve at wrist, ultrasound
mid-arm ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of ulnar nerve, mid-arm, ultrasound
elbow ultrasound | baseline
  Comparison of axial cross-sectional area to Bilateral exploration of ulnar nerve, elbow, ultrasound
ultrasound | Day of the evaluation
  Comparison of axial cross-sectional area to Bilateral exploration of ulnar nerve, mid-forearm, ultrasound
radial nerve ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of radial nerve ultrasound
superficial radial branch nerve ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of superficial radial branch nerve ultrasound
C5, C6 ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of C5, C6 roots ultrasound
sural nerve ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of sural nerve ultrasound
superficial fibular nerve ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of superficial fibular nerve ultrasound
popliteus ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of popliteus tibial nerve at ankle ultrasound
tibial ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of tibial nerveat ankle ultrasound
fibular ultrasound | Baseline
  Comparison of axial cross-sectional area to Bilateral exploration of fibular nerve at the neck ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] El Houjeiry E, Coudray S, Thouvenot E, Ion IM. Spinal cord lesion mimicking a dysimmune myelitis revealing CANVAS syndrome. J Spinal Cord Med. 2023 Mar;46(2):332-336. doi: 10.1080/10790268.2022.2033936. Epub 2022 Mar 2. PMID 35235501